CLINICAL TRIAL: NCT05543044
Title: Examining the Impact of Peer Mentors on Individuals Transitioning to Adult Eating Disorder Treatment: A Feasibility Study
Brief Title: Impact of Peer Mentors on Individuals Transitioning to Adult Eating Disorder Treatment
Acronym: TAY-Mentors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Dr. Aaron Keshen, MD, FRCPC, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1028566
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Peer Mentors; Youth; Feasibility
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAY receiving peer mentor intervention (Experimental): Transition age youth with EDs (n=50) will receive a peer mentor delivered transition intervention
  Interventions: Behavioral: Peer mentor intervention

INTERVENTIONS:
Behavioral: Peer mentor intervention — Peer mentor delivered intervention for transitions to adult-oriented treatment for eating disorders

SUMMARY:
Participants will be males and females aged 16-24 with an eating disorder (ED) diagnosis who are transitioning to adult-oriented ED treatment in Nova Scotia, New Brunswick, or Prince Edward Island. Youth participants will be recruited from community-based clinics, hospital programs, and private practices where ED treatment is delivered. Youth who are interested in participating and provide written consent will be invited to take part in a screening meeting to determine eligibility to participate. Eligible participants will be paired with a peer mentor for a 3-6 month intervention to guide them through the transition to adult-oriented ED treatment. Participants will be asked to complete questionnaire packages before beginning the intervention, after completing the intervention, and 12 months after beginning the intervention. Some youth participants, as well as some of their carers and the peer mentors, will be asked to participate in one-on-one interviews about their experiences with transitions in ED care and the peer mentor intervention. The investigators are conducting this study to determine whether the use of peer mentors is an effective and acceptable means of transition support for youth with EDs. The investigators are also interested in better understanding the experiences of carers and peer mentors who are supporting youth with EDs during their transition in care.

DETAILED DESCRIPTION:
This feasibility study will incorporate quantitative and qualitative methods and utilizes an uncontrolled pretest-posttest quasi-experimental design to examine the effectiveness and acceptability of a peer mentor delivered intervention that aims to improve transitions to adult-oriented care for patients with eating disorders (EDs) aged 16-24.

Youth will be recruited from community-based clinics, hospital programs, and private practices where youth- or adult-oriented ED treatment is delivered across Nova Scotia, New Brunswick, and Prince Edward Island. Clinicians in these settings will be asked to identify potentially eligible youth who will be transitioning to adult-oriented ED care. Potential participants who are interested in participating and provide written consent will meet with a research team member for a screening meeting to determine their eligibility status. Screening will involve the Structured Clinical Interview for DSM-5 Research Version (SCID-5-RV) and the Columbia Suicide Severity Rating Scale (C-SSRS). All screening information will be reviewed by the PI (Dr. Keshen). Participants who are not interested in the study or who fail to meet the eligibility criteria will be given standard options available to treatment age youth.

Youth participants who are found eligible will be connected with a trained peer mentor for a 3-6 month transition intervention. Youth and their peer mentor will meet weekly, bi-weekly, or monthly depending on the phase of the intervention and the needs of the youth. The intervention is divided into 3 phases: phase 1 includes building a sense of trust, rapport, and motivation, as well as the identification of goals, strengths, challenges and barriers related to transition; phase 2 focuses on self-reflection, problem-solving, and transition planning; and phase 3 involves the gradual tapering off and conclusion of the peer mentor relationship.

Youth participants will be asked to complete questionnaire packages before beginning the intervention, after completing the intervention, and 12 months after beginning the intervention. Some youth will also be asked to participate in one-on-one interviews with a research team member at these same time-points. Some youth participants will be asked if they would like to involve a carer in the study, as well. Carers will be invited to participate in a one-on-one interview with a research team member 12 months after the youth they are caring for began the intervention. Peer mentors will be invited to participate in one-on-one interviews at the end of the study. The aim of the interviews is to understand experiences with eating disorder treatment, transitions in care, and the peer mentor intervention.

ELIGIBILITY:
TAY Inclusion Criteria:

* Meets one of the following criteria:

  * 'Aging out' of youth-oriented ED treatment at 19 years-old and unlikely to achieve remission prior to leaving the program (as determined by their clinician[s])
  * Have been deemed incompatible with traditional youth-oriented ED treatment (based on established youth-oriented ED treatment criteria, and determined by their clinician[s])
  * Have requested and/or had a carer request a transition to adult-oriented ED treatment
  * Have been self-referred or referred to adult ED treatment by a clinician (even if they have not been involved in youth-oriented ED treatment)
* Aged 16-24 years old
* Meets criteria for DSM-5 diagnosis of an ED, as confirmed by the Structured Clinical Interview for DSM-5 Research Version (SCID-5-RV)
* Virtually signed informed consent form

TAY Exclusion Criteria:

* Insufficient knowledge of English
* Moderate to high suicide risk rating at screening as assessed by the Columbia Suicide Severity Rating Scale (CSSRS; at the discretion of the PI)

Carer Inclusion Criteria:

* Identified by a TAY participant as a carer
* Aged 18 or older
* Virtually signed informed consent form

Carer Exclusion Criteria:

• Insufficient knowledge of English

PM Inclusion Criteria:

* Certified PM with EDNS
* Providing PM support to TAY study participants
* Virtually signed informed consent form

PM Exclusion Criteria:

• Insufficient knowledge of English

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Autonomous Motivation | Baseline, 3-6 months, 12 months
  This will be measured at Baseline, Post-Intervention, and 12-Month Follow-Up, using The Treatment Self-Regulation Questionnaire (TSRQ; Levesque et al., 2007). The TSRQ is a reliable and valid self-report questionnaire that assesses the type of motivation patients use (autonomous or external/controlled) when engaging in a health behaviour or treatment. The TSRQ consists of 12 questions with scores ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The TSRQ can be modified to measure specific health care outcomes (e.g., ED related). Further, the TSRQ has previously been used to detect changes in autonomous motivation before and after health-related interventions, including over six-month timeframes (e.g., Stamp et al., 2016; Knittle et al., 2015). A recent scoping review determined that there are no validated quantitative measures for specifically evaluating mental health related transition interventions for TAY (Cleverly et al., 2018).

SECONDARY OUTCOMES:
Completed Transitions | 12 months
  Engagement in adult-oriented service could include: a) one session (or more) of individual psychotherapy aimed at treating the ED (as determined by the PI); b) an admission into AEDP (i.e., group-based Day Program or Inpatient); and c) the youth is on the wait-list to start adult treatment. Initiation of adult services can be through referral from any clinician or self-referral. Although our measurement of a completed transition is a dichotomous variable, we will also collect exploratory data to examine the degree of service uptake in the adult-oriented treatment (low, medium, and high use as defined by McClelland et al., 2020). This will allow us to explore not only whether the youth transitioned or not, but also to what degree they engaged in an adult service after the transition.
Patient acceptability | Throughout study completion, 12 months
  This will be measured at Baseline, Post-Intervention, and 12-Month Follow-Up, using the Health Care Climate Questionnaire (HCCQ; Williams, et al., 1996) at Baseline, Post-Intervention, and 12-Month Follow-Up. The HCCQ measures the extent to which patients feel that providers take full account of their perspective, offer choice and information, encourage self-initiation, provide rationale, and accept patient decisions. The HCCQ is a companion scale to the TSRQ, and has been positively associated with autonomous motivation and treatment adherence (Williams et al., 2006; Chan et al., 2009). The HCCQ is a valid and reliable 6-item self-report questionnaire with scores ranging from 1 ("strongly disagree") to 7 ("strongly agree").

OTHER OUTCOMES:
Change in eating disorder symptomatology | Baseline, 3-6 months, 12 months
  This will be measured at Baseline, Post-Intervention, and 12-Month Follow-Up, using the Eating Disorder Examination Questionnaire (EDE-Q; Fairburn & Beglin, 1994), a validated and reliable 28-item self-report questionnaire.
Change in clinical impairment | Baseline, 3-6 months, 12 months
  This will be measured at Baseline, Post-Intervention, and 12-Month Follow-Up, using the Clinical Impairment Assessment (CIA; Bohn & Fairburn, 2008), which is a reliable and validated 16-item self-report questionnaire that measures functional impairment over the last 28 days. Higher scores on the CIA indicate more impairment.
Change in feelings of competence about participating in eating disorder treatment | Baseline, 3-6 months, 12 months
  This will be measured at Baseline, Post-Intervention, and 12-Month Follow-Up using the Perceived Competence Scale (PCS; Williams et al., 1995), a companion scale in a questionnaire package that includes the TSRQ. The PCS is a valid and reliable tool that evaluates feelings of competence about participating in a health behaviour or treatment. The PCS is a 4-item self-report questionnaire with scores ranging from 1 ("not at all true") to 7 ("very true").

CONTACTS AND LOCATIONS:
Overall Officials: Aaron K Keshen, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Abbie J Lane Memorial Building - QEII, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Austin A, Flynn M, Richards K, Hodsoll J, Duarte TA, Robinson P, Kelly J, Schmidt U. Duration of untreated eating disorder and relationship to outcomes: A systematic review of the literature. Eur Eat Disord Rev. 2021 May;29(3):329-345. doi: 10.1002/erv.2745. Epub 2020 Jun 23. PMID 32578311
- [Background] Beveridge J, Phillipou A, Jenkins Z, Newton R, Brennan L, Hanly F, Torrens-Witherow B, Warren N, Edwards K, Castle D. Peer mentoring for eating disorders: results from the evaluation of a pilot program. J Eat Disord. 2019 Jun 3;7:13. doi: 10.1186/s40337-019-0245-3. eCollection 2019. PMID 31171969
- [Background] Bohn, K., & Fairburn, C. G. (2008). The clinical impairment assessment questionnaire (CIA). Cognitive behavioral therapy for eating disorders, 1-3
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3, 77-101. doi:10.1191/1478088706qp063oa
- [Background] Broad, B. (1999). Improving the health of children and young people leaving care. Adoption & Fostering, 23(1), 40-48
- [Background] Burke NL, Schaefer LM, Hazzard VM, Rodgers RF. Where identities converge: The importance of intersectionality in eating disorders research. Int J Eat Disord. 2020 Oct;53(10):1605-1609. doi: 10.1002/eat.23371. Epub 2020 Aug 28. PMID 32856342
- [Background] Clausen L, Lubeck M, Jones A. Motivation to change in the eating disorders: a systematic review. Int J Eat Disord. 2013 Dec;46(8):755-63. doi: 10.1002/eat.22156. Epub 2013 Jul 11. PMID 23847134
- [Background] Cleverley K, Rowland E, Bennett K, Jeffs L, Gore D. Identifying core components and indicators of successful transitions from child to adult mental health services: a scoping review. Eur Child Adolesc Psychiatry. 2020 Feb;29(2):107-121. doi: 10.1007/s00787-018-1213-1. Epub 2018 Oct 8. PMID 30294756
- [Background] Research design: qualitative, quantitative and mixed methods approaches Research design: qualitative, quantitative and mixed methods approaches Creswell John W Sage 320 pound29 0761924426 0761924426 [Formula: see text]. Nurse Res. 2004 Sep 1;12(1):82-83. doi: 10.7748/nr.12.1.82.s2. PMID 28718745
- [Background] Crocker, C., Cox, A., Abidi, S., Ursuliak, Z., Epstein, N., Hughes, J., Crown, M. & Tibbo, P. (2020). M238. Creation Of A Peer Support Program To Support Transitions In Care From Early Intervention Services For Psychosis. Schizophrenia Bulletin, 46(Supplement_1), S226-S226.
- [Background] Culbert KM, Racine SE, Klump KL. Research Review: What we have learned about the causes of eating disorders - a synthesis of sociocultural, psychological, and biological research. J Child Psychol Psychiatry. 2015 Nov;56(11):1141-64. doi: 10.1111/jcpp.12441. Epub 2015 Jun 19. PMID 26095891
- [Background] Deci, E., & Ryan, R. M. (1985). Intrinsic motivation and self-determination in human behavior. Springer Science & Business Media.
- [Background] Dimitropoulos G, Toulany A, Herschman J, Kovacs A, Steinegger C, Bardsley J, Sandhu S, Gregory C, Colton P, Anderson J, Kaufman M. A qualitative study on the experiences of young adults with eating disorders transferring from pediatric to adult care. Eat Disord. 2015;23(2):144-62. doi: 10.1080/10640266.2014.976106. Epub 2014 Nov 17. PMID 25402167
- [Background] Dimitropoulos G, Tran AF, Agarwal P, Sheffield B, Woodside B. Navigating the transition from pediatric to adult eating disorder programs: perspectives of service providers. Int J Eat Disord. 2012 Sep;45(6):759-67. doi: 10.1002/eat.22017. Epub 2012 Mar 19. PMID 22431280
- [Background] Dimitropoulos G, Tran AF, Agarwal P, Sheffield B, Woodside B. Challenges in making the transition between pediatric and adult eating disorder programs: a qualitative study from the perspective of service providers. Eat Disord. 2013;21(1):1-15. doi: 10.1080/10640266.2013.741964. PMID 23241086
- [Background] Embrett MG, Randall GE, Longo CJ, Nguyen T, Mulvale G. Effectiveness of Health System Services and Programs for Youth to Adult Transitions in Mental Health Care: A Systematic Review of Academic Literature. Adm Policy Ment Health. 2016 Mar;43(2):259-69. doi: 10.1007/s10488-015-0638-9. PMID 25708229
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Gilmer TP, Ojeda VD, Leich J, Heller R, Garcia P, Palinkas LA. Assessing needs for mental health and other services among transition-age youths, parents, and providers. Psychiatr Serv. 2012 Apr;63(4):338-42. doi: 10.1176/appi.ps.201000545. PMID 22337004
- [Background] Gopalan G, Lee SJ, Harris R, Acri MC, Munson MR. Utilization of peers in services for youth with emotional and behavioral challenges: A scoping review. J Adolesc. 2017 Feb;55:88-115. doi: 10.1016/j.adolescence.2016.12.011. Epub 2017 Jan 7. PMID 28068538
- [Background] le Grange D. Family therapy for adolescent anorexia nervosa. J Clin Psychol. 1999 Jun;55(6):727-39. doi: 10.1002/(sici)1097-4679(199906)55:63.0.co;2-3. PMID 10445863
- [Background] Griffiths S, Mond JM, Murray SB, Touyz S. The prevalence and adverse associations of stigmatization in people with eating disorders. Int J Eat Disord. 2015 Sep;48(6):767-74. doi: 10.1002/eat.22353. Epub 2014 Sep 5. PMID 25196068
- [Background] Guss CE, Williams DN, Reisner SL, Austin SB, Katz-Wise SL. Disordered Weight Management Behaviors, Nonprescription Steroid Use, and Weight Perception in Transgender Youth. J Adolesc Health. 2017 Jan;60(1):17-22. doi: 10.1016/j.jadohealth.2016.08.027. Epub 2016 Oct 28. PMID 28029539
- [Background] Hanly F, Torrens-Witherow B, Warren N, Castle D, Phillipou A, Beveridge J, Jenkins Z, Newton R, Brennan L. Peer mentoring for individuals with an eating disorder: a qualitative evaluation of a pilot program. J Eat Disord. 2020 Jul 1;8:29. doi: 10.1186/s40337-020-00301-8. eCollection 2020. PMID 32626579
- [Background] Hoek HW. Incidence, prevalence and mortality of anorexia nervosa and other eating disorders. Curr Opin Psychiatry. 2006 Jul;19(4):389-94. doi: 10.1097/01.yco.0000228759.95237.78. PMID 16721169
- [Background] Jones BA, Haycraft E, Bouman WP, Brewin N, Claes L, Arcelus J. Risk Factors for Eating Disorder Psychopathology within the Treatment Seeking Transgender Population: The Role of Cross-Sex Hormone Treatment. Eur Eat Disord Rev. 2018 Mar;26(2):120-128. doi: 10.1002/erv.2576. Epub 2018 Jan 10. PMID 29318711
- [Background] Mahon, J. (2000). Dropping out from psychological treatment for eating disorders: What are the issues?. European Eating Disorders Review: the Professional Journal of the Eating Disorders Association, 8(3), 198-216. https://doi.org/10.1002/(SICI)1099-0968(200005)8:3%3C198::AID-ERV356%3E3.0.CO;2-3
- [Background] McClelland J, Simic M, Schmidt U, Koskina A, Stewart C. Defining and predicting service utilisation in young adulthood following childhood treatment of an eating disorder. BJPsych Open. 2020 Apr 6;6(3):e37. doi: 10.1192/bjo.2020.13. PMID 32248870
- [Background] McClelland J, Hodsoll J, Brown A, Lang K, Boysen E, Flynn M, Mountford VA, Glennon D, Schmidt U. A pilot evaluation of a novel First Episode and Rapid Early Intervention service for Eating Disorders (FREED). Eur Eat Disord Rev. 2018 Mar;26(2):129-140. doi: 10.1002/erv.2579. PMID 29460477
- [Background] Munoz-Solomando A, Townley M, Williams R. Improving transitions for young people who move from child and adolescent mental health services to mental health services for adults: lessons from research and young people's and practitioners' experiences. Curr Opin Psychiatry. 2010 Jul;23(4):311-7. doi: 10.1097/YCO.0b013e32833a51e2. PMID 20520550
- [Background] Murray SB, Nagata JM, Griffiths S, Calzo JP, Brown TA, Mitchison D, Blashill AJ, Mond JM. The enigma of male eating disorders: A critical review and synthesis. Clin Psychol Rev. 2017 Nov;57:1-11. doi: 10.1016/j.cpr.2017.08.001. Epub 2017 Aug 2. PMID 28800416
- [Background] Murray SB. Gender Identity and Eating Disorders: The Need to Delineate Novel Pathways for Eating Disorder Symptomatology. J Adolesc Health. 2017 Jan;60(1):1-2. doi: 10.1016/j.jadohealth.2016.10.004. Epub 2016 Nov 10. No abstract available. PMID 27838236
- [Background] Pottick KJ, Bilder S, Vander Stoep A, Warner LA, Alvarez MF. US patterns of mental health service utilization for transition-age youth and young adults. J Behav Health Serv Res. 2008 Oct;35(4):373-89. doi: 10.1007/s11414-007-9080-4. Epub 2007 Nov 17. PMID 18026842
- [Background] Sansfacon J, Gauvin L, Fletcher E, Cottier D, Rossi E, Kahan E, Israel M, Steiger H. Prognostic value of autonomous and controlled motivation in outpatient eating-disorder treatment. Int J Eat Disord. 2018 Oct;51(10):1194-1200. doi: 10.1002/eat.22901. Epub 2018 Sep 1. PMID 30171769
- [Background] Singh SP, Paul M, Ford T, Kramer T, Weaver T, McLaren S, Hovish K, Islam Z, Belling R, White S. Process, outcome and experience of transition from child to adult mental healthcare: multiperspective study. Br J Psychiatry. 2010 Oct;197(4):305-12. doi: 10.1192/bjp.bp.109.075135. PMID 20884954
- [Background] Strauss, A., & Corbin, J. (1998). Basics of qualitative research: Procedures and techniques for developing grounded theory.
- [Background] Steiger H, Sansfacon J, Thaler L, Leonard N, Cottier D, Kahan E, Fletcher E, Rossi E, Israel M, Gauvin L. Autonomy support and autonomous motivation in the outpatient treatment of adults with an eating disorder. Int J Eat Disord. 2017 Sep;50(9):1058-1066. doi: 10.1002/eat.22734. Epub 2017 Jun 14. PMID 28842966
- [Background] Thapliyal P, Hay P, Conti J. Role of gender in the treatment experiences of people with an eating disorder: a metasynthesis. J Eat Disord. 2018 Aug 13;6:18. doi: 10.1186/s40337-018-0207-1. eCollection 2018. PMID 30123504
- [Background] Thomas, D. R. (2006). A general inductive approach for analyzing qualitative evaluation data. American Journal of Evaluation, 27(2), 237-246.
- [Background] Treasure J, Schmidt U, Hugo P. Mind the gap: service transition and interface problems for patients with eating disorders. Br J Psychiatry. 2005 Nov;187:398-400. doi: 10.1192/bjp.187.5.398. PMID 16260812
- [Background] Wagner R, Stevens JR. Clinical Barriers to Effective Treatment of Eating Disorders and Co-occurring Psychiatric Disorders in Transgendered Individuals. J Psychiatr Pract. 2017 Jul;23(4):284-289. doi: 10.1097/PRA.0000000000000248. PMID 28749833
- [Background] Williams, G. C., Gagné, M., Ryan, R. M., & Deci, E. L. (1999). Supporting autonomy to motivate smoking cessation: A test of self-determination theory. Unpublished manuscript, University of Rochester, New York.
- [Background] Winston AP, Paul M, Juanola-Borrat Y. The same but different? Treatment of anorexia nervosa in adolescents and adults. Eur Eat Disord Rev. 2012 Mar;20(2):89-93. doi: 10.1002/erv.1137. Epub 2011 Sep 13. PMID 21913286